CLINICAL TRIAL: NCT00889512
Title: The Luveris® In Vitro Fertilization Trial: The Effect of Recombinant Luteinizing Hormone on Follicular Response, Oocyte Quality, and Pregnancy in In-Vitro Fertilization Treatment Cycles in Women Without Endogenous LH Activity.
Brief Title: The Luveris In Vitro Fertilization Trial
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Drug no longer available by manufacturer
Sponsor: University Reproductive Associates (Other)
Collaborators: EMD Serono (Industry)
Responsible Party: Principal Investigator, Peter McGovern, MD, Director, University Reproductive Associates
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0120080358
Record Dates: First submitted 2009-04-28; First posted 2009-04-29 (Estimated); Results first posted 2014-10-23 (Estimated); Last update posted 2018-08-07 (Actual); Status verified 2018-07

CONDITIONS: Infertility; Hypothalamic Amenorrhea; Hyperprolactinemia
MeSH Terms: conditions — Infertility; Hyperprolactinemia | interventions — Luteinizing Hormone, beta Subunit

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Luveris Fixed dose (Active Comparator): Participants in this arm will take Gonal F® and the same dose of Luveris® throughout the cycle. Their dose of Gonal F® will be adjusted throughout the cycle based on their response to the medication. The Luveris® dose will remain constant throughout.
  Interventions: Drug: Luveris fixed dose
- Luveris increasing dose (Experimental): Patients assigned to this group will gradually reduce the Gonal F® dose while increasing the Luveris® dose during the cycle, which more closely mimics the natural menstrual cycle.
  Interventions: Drug: Luveris increasing dose

INTERVENTIONS:
Drug: Luveris fixed dose — Luveris 75IU daily throughout ovarian stimulation
  Arms: Luveris Fixed dose
Drug: Luveris increasing dose — Luveris 75IU until estradiol level reaches 250 pg/ml then increasing to 75IU BID for two days, then TID until hCG
  Arms: Luveris increasing dose

SUMMARY:
The purpose of this study is to develop a new protocol using two different types of fertility drugs that is more similar to the way the hormones act in a normal menstrual cycle (period).

We are recruiting women who are trying to get pregnant through In Vitro Fertilization (IVF) who either have a high prolactin level (a hormone normally found in your blood that is produced in the brain) or have a condition known as hypothalamic amenorrhea in which one does not get regular periods due to low hormone levels.

The ovaries can be stimulated with Follicle Stimulating Hormone (FSH) alone and with FSH and Luteinizing Hormone (LH). FSH causes eggs to be made while LH causes estrogen (hormone) production. The women in this study have low hormone levels and need both FSH and LH. Luveris® (LH hormone) is a new drug approved for egg production and is used in IVF. There is no set amount of LH nor a set protocol for LH use. Therefore, we are testing this new regimen. One group of women will receive a fixed dose of LH throughout their cycle while the other will decrease the dose of FSH while at the same time increasing the LH dose which is what happens in the natural menstrual cycle.

ELIGIBILITY:
Inclusion Criteria:

1. 30 women under 38 years old at time of signing Informed Consent Form.
2. Evidence of hypothalamic amenorrhea (irregular menses and FSH and LH <5 mIU/mL), uncorrected hyperprolactinemia (prolactin levels 10% above the upper limit of normal) or iatrogenic hypothalamic hypogonadism secondary to GnRHa suppression.
3. In good general health off of current medications which may confound response to study medications except GnRHa (Lupron Depot).
4. Desire to seek pregnancy actively during the study period.
5. A normal uterine cavity must have been confirmed by either hysteroscopy or hydrosonogram within two years of entering the study.
6. A semen analysis on the male partner deemed adequate for IVF by the attending physician within the past year or donor sperm available for insemination.
7. Only one treatment cycle per patient will be studied.

Exclusion Criteria:

1. uncorrected thyroid disease.
2. heart disease (New York Heart Association Class II or higher).
3. a history of, or suspected cervical, endometrial, or breast cancer. A normal Pap smear result within the last 24 months will be required.
4. enrolled into other studies that require medications, limit sex, or otherwise prevent compliance with the protocol at the same time.
5. to take other medications known to affect reproduction.

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2009-04 (Actual); Primary Completion 2013-05 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University Reproductive Associates, Hasbrouck Heights, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Luveris Fixed Dose | Luveris Increasing Dose
Started | 5 | 9
Completed | 5 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Luveris Fixed Dose | Luveris Increasing Dose | Total
Number analyzed (Participants) | 5 | 9 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 9 | 14
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 9 | 14
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: The Primary Outcome Will be Number of Large Follicles (16 mm or Greater in Diameter) and Midsize Follicles (Greater Than 12mm But Less Than 16mm) in Both Groups on the Day of Meeting Size Criteria for hCG.
Time Frame: 2 years
Measure: Median (Full Range); unit: number of follicles
Arm/Group | Luveris Fixed Dose | Luveris Increasing Dose
Number analyzed (Participants) | 5 | 9
number of follicles
  Large Follicles | 3 [3 to 6] | 3 [2 to 5]
  Midsize Follicles | 4 [2 to 10] | 4 [1 to 8]

ADVERSE EVENTS:
Time Frame: 1 year
Description: No adverse or serious adverse events occurred
Groups:
- Group A: Participants in this arm will take Gonal F® and the same dose of Luveris® throughout the cycle. Their dose of Gonal F® will be adjusted throughout the cycle based on their response to the medication. The Luveris® dose will remain constant throughout.
  Luveris fixed dose: Luveris 75IU daily throughout ovarian stimulation
- Group B: Patients assigned to this group will gradually reduce the Gonal F® dose while increasing the Luveris® dose during the cycle, which more closely mimics the natural menstrual cycle.
  Luveris increasing dose: Luveris 75IU until estradiol level reaches 250 pg/ml then increasing to 75IU BID for two days, then TID until hCG
Arm/Group | Group A | Group B
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/9
Other Adverse Events (participants affected / at risk) | 0/5 | 0/9

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed;

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No